CLINICAL TRIAL: NCT00225758
Title: Lapatinib in Endocrine-Resistant Metastatic Breast Cancer
Brief Title: Lapatinib in Metastatic Breast Cancer Resistant to Hormone Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Gary Schwartz (Other)
Collaborators: University of Colorado, Denver (Other); North Shore University Hospital (Other)
Responsible Party: Sponsor-Investigator, Gary Schwartz, Staff Physician, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-0520
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Metastatic Breast Cancer
Keywords: breast cancer; endocrine therapy; drug resistance; lapatinib; epidermal growth factor receptor
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Subjects will continue on their prior endocrine therapy with the addition of lapatinib at 1500 mg once daily for 26 weeks or longer.
  Interventions: Drug: Lapatinib

INTERVENTIONS:
Drug: Lapatinib — 1500 mg po daily for 26 weeks or longer
  Other Names: Tykerb

SUMMARY:
Two thirds or more of breast cancers are dependent on estrogen for growth. We use a number of estrogen-blocking medicines for treatment of metastatic breast cancer. The treatment response to these agents is unpredictable, however, and approximately one-third of patients with metastatic breast cancer with receptors for estrogen or progesterone have no benefit from hormonal therapy. Nearly all patients with metastatic breast cancer will eventually become resistant to hormonal therapy despite the fact that the hormone receptors are still present.

Some cells make a different class of growth factor receptor called the Epidermal Growth Factor Receptor. There is a growing body of experimental evidence showing that breast cancer cells that make Epidermal Growth Factor Receptors are more resistant to hormonal therapy and have a poorer prognosis. Several investigators have found that the Epidermal Growth Factor Receptor can activate the estrogen receptor, even in the presence of estrogen-blocking drugs. Growth of these cells can be slowed by blockade of both Epidermal Growth Factor Receptor signaling and estrogen-receptor signaling. Lapatinib is a small molecule which can inhibit two different forms of the Epidermal Growth Factor Receptor. It has been studied in people with a number of different cancers, including breast cancer, and a safe dose and its common side effects have been defined.

Our hypothesis is that the Epidermal Growth Factor Receptor is the dominant receptor pathway used by breast cancers in our patients with hormone-resistant tumors. Drugs like lapatinib which block several forms of the Epidermal Growth Factor Receptor would best be able to reverse resistance to hormonal agents.

DETAILED DESCRIPTION:
All patients must have stopped their endocrine two to four weeks or longer prior to entry on study. Upon enrollment, patients will begin lapatinib at 1500 mg once a day orally. The original endocrine therapy will resume two weeks later. The lapatinib will be continued for a maximum of 26 weeks.

A history, physical examination, blood counts, and chemistries will be done at baseline, and at regular intervals through the course of the study. A CT scan and bone scan will be done prior to treatment and at weeks 14 and 26. Assays for plasma DNA will be performed on blood sampled at baseline and at multiple time points throughout the course of treatment. Percutaneous biopsies will be taken in selected patients with accessible disease, 72 hours or less prior to the start of lapatinib, and again 13-15 days, and 27-29 days following the start of lapatinib. The day 13-15 biopsy will be done just prior to the resumption of the patient's endocrine therapy. Assays for phospho-ERK, phospho-Akt, Cyclin D1, Ki-67, and IRS-1 will be performed by conventional immunohistochemistry on the biopsied tissue.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically proven metastatic breast cancer.
* Patients with either estrogen or progesterone receptor positivity on the most recently examined tumor biopsy.
* Patients must have most recently been using an anti-estrogen (tamoxifen, toremifene, raloxifene, or fulvestrant) or an aromatase inhibitor.
* Patients must have had either a partial response or better, or stable disease for 24 weeks or longer, followed by disease progression, on the current or most recent hormonal therapy for management of metastatic breast cancer.
* Patients must be enrolled within six weeks of defining disease progression on hormonal therapy.
* Patients must have stopped fulvestrant at least four weeks prior and other endocrine therapy at least two weeks prior to enrollment on study.
* Patients must have either measurable disease or at least one evaluable bone lesion that has not been irradiated. Measurable disease is not necessary.
* Estimated life expectancy of at least 6 months.
* ECOG performance status 0-2.
* Adequate hematologic, hepatic, and renal function.
* Patients must be post-menopausal, or they must be practicing either abstinence or an adequate method of contraception, or their sexual partner must be sterile.
* All patients must be able to swallow, retain, and absorb oral medications.
* All patients must be able to give informed consent indicating that they are aware of the investigational nature of this study.

Exclusion Criteria:

* Patients may not have received an investigational agent within the prior four weeks.
* Patients may not have received trastuzumab within three weeks of study entry.
* Patients may not have had major surgery within the prior two weeks.
* Patients may not have Class III or IV heart failure as defined by the NYHA functional classification system.
* Patients may not have a left ventricular ejection fraction < 40% based on MUGA or echocardiogram.
* Patients may not have uncontrolled brain metastases or leptomeningeal disease.
* Patients may not have rapidly progressive visceral metastases.
* Patients may not have a serious illness or conditions including clinically significant cardiac disease, angina pectoris, serious psychiatric disorder, or an active infection.
* Patients may not be receiving concurrent medications (listed in the protocol) which may interact with lapatinib during treatment with lapatinib.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary N Schwartz, MD, Principal Investigator — Norris Cotton Cancer Center
Locations (3):
- United States (3):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - North Shore University Hospital, Lake Success, New York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects will continue on the same endocrine therapy they had been taking at the time of disease progression.
Groups:
- Endocrine Therapy Plus Lapatinib: Subjects will continue on their prior endocrine therapy with the addition of lapatinib at 1500 mg once daily for 26 weeks or longer.
  Lapatinib: 1500 mg po daily for 26 weeks or longer
Period: Overall Study
Arm/Group | Endocrine Therapy Plus Lapatinib
Started | 27
Completed | 23
Not Completed | 4
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Arm/Group | Endocrine Therapy Plus Lapatinib
Number analyzed (Participants) | 27
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [52 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Determine the Response Rate and Progression Free Survival of Hormone Therapy-resistant Patients With Metastatic Breast Cancer Treated With the Same Continued Hormonal Agent With the Addition of Lapatinib.
Description: A response is defined as stable disease or better at 26 weeks. Twenty two patients are evaluable for response
Time Frame: 26 weeks
Population: Of the 27 enrolled subjects, five subjects came off study due to toxicity prior to week 14, at the time of the first restaging. The remaining 22 subjects are evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Endocrine Therapy Plus Lapatinib
Number analyzed (Participants) | 22
Participants | 8

2. Primary Outcome: Progression-free Survival
Description: Progression-free survival is the time between date on study and progression based on RECIST criteria.
Time Frame: Up to 575 days
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Lapatinib Plus Endocrine Therapy: Subjects receive lapatinib 1500 mg daily in addition to their prior endocrine therapy.
Arm/Group | Lapatinib Plus Endocrine Therapy
Number analyzed (Participants) | 22
days | 150 [95 to 300]

3. Secondary Outcome: Determine the Toxicities of the Combination of the Hormonal Agent and Lapatinib in Patients With Metastatic Breast Cancer
Time Frame: 26 weeks
Population: All 27 subjects are evaluable for toxicity
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib Plus Endocrine Therapy
Number analyzed (Participants) | 27
Participants
  Severe adverse events: Subjects with the adverse event | 0
  Severe adverse events: Subjects without the adverse event | 27
  Adverse events with a frequency of 5% or more: Subjects with the adverse event | 23
  Adverse events with a frequency of 5% or more: Subjects without the adverse event | 4

4. Secondary Outcome: Determine Changes in Activation of Tumor Cell ERK and Akt, as Between the Hormonal Agent and Lapatinib Contributes to the Molecular Pharmacodynamic Effect Postulated Above.
Time Frame: 4 weeks
Population: None of the patients had the recommended biopsies done as the biopsies were optional, and over half the patients had either bone-only disease or only non-biopsiable soft tissue disease.
Groups:
- Lapatinib Plus Prior Endocrine Therapy: Subjects will continue on their prior endocrine therapy with the addition of lapatinib at 1500 mg once daily for 26 weeks or longer.
  Lapatinib: 1500 mg po daily for 26 weeks or longer
Arm/Group | Lapatinib Plus Prior Endocrine Therapy
Number analyzed (Participants) | 0

5. Secondary Outcome: Determine Whether Changes in Plasma DNA Concentrations Are Predictive Markers of an Early Response to Lapatinib
Time Frame: 14 weeks
Population: Plasma DNA assays were not done due to difficulty obtaining plasma specimens from the outside sites, and technical problems with the assay in the specimens collected at our institution..
Arm/Group | Lapatinib Plus Prior Endocrine Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Lapatinib Plus Endocrine Therapy
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 23/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lapatinib Plus Endocrine Therapy (N=27)
Grade 3 diarrhea (Gastrointestinal disorders) | 5 (8)
Grade 2 diarrhea (Gastrointestinal disorders) | 12 (21)
Grade 3 cellulitis (Infections and infestations) | 3 (3)
Grade 3 hypokalemia (Blood and lymphatic system disorders) | 3 (3)
Grade 2 anemia (Blood and lymphatic system disorders) | 3 (3)
Grade 2 vomiting (Gastrointestinal disorders) | 2 (4)
Grade 2 nausea (Gastrointestinal disorders) | 2 (3)
Grade 2 lymphopenia (Investigations) | 5 (7)
Grade 2 fatigue (General disorders) | 5 (5)
Grade 2 rash (Skin and subcutaneous tissue disorders) | 3 (4)
Grade 2 weight loss (Metabolism and nutrition disorders) | 2 (2)
Grade 2 skeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Grade 2 edema (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No